CLINICAL TRIAL: NCT01043029
Title: Effects of 150 mcg Aleglitazar on Renal Function in Patients With Type 2 Diabetes and Moderate Renal Impairment, as Compared to Actos®
Brief Title: A Study of Aleglitazar in Type 2 Diabetes Patients With Moderate Renal Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC22419; 2009-012270-12
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — aleglitazar; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- aleglitazar (Experimental)
  Interventions: Drug: aleglitazar
- pioglitazone (Active Comparator)
  Interventions: Drug: pioglitazone

INTERVENTIONS:
Drug: aleglitazar — Aleglitazar 150 mcg po daily for 52 weeks
  Arms: aleglitazar
Drug: pioglitazone — Pioglitazone 45 mg po daily for 52 weeks
  Arms: pioglitazone

SUMMARY:
This multi-center, randomized, double-blind, active controlled, parallel-group study in type 2 diabetes patients with moderate renal impairment will evaluate the effect on renal function and the safety and tolerability of aleglitazar compared with pioglitazone. Patients will be randomized to receive either 150 mcg aleglitazar or 45 mg pioglitazone as daily oral doses. In addition, a diet and exercise plan will also be implemented during the anticipated time on study treatment of 52 weeks. The target sample size is 200-400 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >/= 18 years of age
* Diabetes mellitus, Type 2
* Moderately impaired kidney function
* Drug naive or up to 2 antihyperglycemic medications at stable dose for over 1 month at screening
* BMI 25-35

Exclusion Criteria:

* Current or previous treatment with a thiazolidinedione
* Current or previous treatment with insulin
* Treatment with fibrates <3 months prior to screening
* History of renal disease other than diabetic nephropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2010-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Renal function: estimated glomerular filtration rate | Week 60

SECONDARY OUTCOMES:
Safety, Tolerability: Adverse events (AEs), laboratory parameters | AEs: Throughout study, laboratory assessments: Week 2, 4, 8, 12, 16, 20, 26, 39, 52, 56, 60
Renal function: estimated glomerular filtration rate | Week 52
Effect on blood hemoglobin | Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (66):
- Australia (7):
  - Camperdown, New South Wales
  - St Leonards, New South Wales
  - Brisbane, Queensland
  - Elizabeth Vale, South Australia
  - Richmond, South Australia
  - Launceston, Tasmania
  - Melbourne, Victoria
- Brazil (3):
  - Fortaleza, Ceará
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
- Colombia (4):
  - Barranquilla
  - Bogotá
  - Bucaramanga
  - Medellin-Antioquia
- San Salvador, El Salvador
- Germany (13):
  - Aschaffenburg
  - Berlin
  - Damme
  - Dresden
  - Essen
  - Falkensee
  - Mainz
  - Münster
  - Neuwied
  - Reichenbach
  - Rostock
  - Sulzbach-Rosenberg
  - Würzburg
- Hong Kong (2):
  - Hong Kong
  - Tuenmen
- Hungary (8):
  - Baja
  - Budapest
  - Debrecen
  - Kecskemét
  - Miskolc
  - Sátoraljaújhely
  - Szeged
  - Szekszárd
- Italy (5):
  - Genoa, Liguria
  - Bergamo, Lombardy
  - Cusano Milanino, Lombardy
  - Milan, Lombardy
  - Pavia, Lombardy
- Mexico (6):
  - Aguascaliente
  - Chihuahua City
  - Cuernavaca
  - Durango
  - Guadalajara
  - Pachuca
- Peru (2):
  - Arequipa
  - Lima
- Romania (6):
  - Bucharest
  - Cluj-Napoca
  - Iași
  - Ploieşti
  - Sibiu
  - Târgu Mureş
- Russia (5):
  - Chelyabinsk
  - Moscow
  - Saint Petersburg
  - Saratov
  - Yaroslavl
- Slovakia (4):
  - Bratislava
  - Dolný Kubín
  - Levice
  - Lučenec

REFERENCES:
- [Derived] Ruilope L, Hanefeld M, Lincoff AM, Viberti G, Meyer-Reigner S, Mudie N, Wieczorek Kirk D, Malmberg K, Herz M. Effects of the dual peroxisome proliferator-activated receptor-alpha/gamma agonist aleglitazar on renal function in patients with stage 3 chronic kidney disease and type 2 diabetes: a Phase IIb, randomized study. BMC Nephrol. 2014 Nov 18;15:180. doi: 10.1186/1471-2369-15-180. PMID 25407798